CLINICAL TRIAL: NCT06150222
Title: Retrospective Cervical Cancer Oligo States (Recurrence, Metastasis) Multicentre Outcomes Study (Retro-COSMOS). An EMBRACE Collaborative Initiative in Recurrent and Metastatic Cervix Cancer.
Brief Title: Retrospective Cervical Cancer Oligo States (Recurrence, Metastasis) Multicentre Outcomes Study
Acronym: Retro-COSMOS
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Prof. Dr. Remi A. Nout, Head of Department of Radiation Oncology, Erasmus Medical Center
Other Study IDs: MEC-2022-0355/ TMC-IEC-900891
Record Dates: First submitted 2023-09-29; First posted 2023-11-29 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Cancer, Cervical; Recurrence; Metastasis
Keywords: Reirradiation; OligoRecurrence; Oligometastasis
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Concurrent Chemoradiation, Systemic Chemotherapy other locally directed therapies (like surgery, ablation, etc.) — The aim is to include all patients with (induced) oligo metastatic and oligo recurrent settings, irrespective of whether treated with concurrent chemoradiation, systemic chemotherapy, or with other locally directed therapies (like surgery, ablation, etc.)

SUMMARY:
This multi centric international retrospective study aims to register patients with oligo metastatic and oligo recurrent cervical cancer. The study will register patients in planned period with an aim to analyse clinical outcomes with or without use of radiation in this setting.

DETAILED DESCRIPTION:
Detailed clinical protocol can be obtained by contacting the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical cancer with (induced) oligo-metastatic and/or oligo-recurrent cervix cancer whether treated or not treated with radiation. These patients may have received previous treatment within or outside approved clinical trials/studies.
2. Patients with poly-metastatic disease with good response to systemic chemotherapy and treated with radiation to recurrence or metastatic site.
3. Patients treated with radical doses at the time of first diagnosis of oligo-metastasis/oligo-recurrence and present with further oligo-progression.
4. Patients with oligo-metastasis or oligo-recurrence treated with other locally directed therapies (like surgery, ablation, etc.) are also permitted.

Exclusion Criteria:

1. Gynecological cancer other than cervical cancer
2. Persistent Poly-metastatic disease post systemic treatment
3. Receiving investigational new drugs at the time of relapse as part of other ongoing trials
4. No clinical follow up after treatment

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with (induced) oligo metastatic and oligo recurrent settings irrespective of whether radiation was used or not.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | From date of diagnosis of recurrence untill the date of death due to any cause or date of censoring at the last time the subject was known to be alive, whichever came first, assessed upto 3 years after initiation of the study
  To estimate overall survival of patients diagnosed with oligo-recurrent and (induced) oligo-metastatic cervix cancer.

SECONDARY OUTCOMES:
3-year Infield progression free survival | From date of first disease progression to date of subsequent progression or death from any cause, whichever came first, assessed upto 3 years after initiation of the study
  To estimate infield progression-free survival and progression-free interval of patients diagnosed with oligo-recurrent and (induced) oligo-metastatic cervix cancer.
3- year Progression free survival | From date of first disease progression to subsequent disease progression or death from any cause, whichever came first, assessed upto 3 years after initiation of the study
  To estimate overall progression-free survival of patients diagnosed with oligo-recurrent and (induced) oligo-metastatic cervix cancer.
Dose response relationship of nodal and visceral progressions | From date of start of treatment of disease progression, assessed upto 3 years
  Radiation Dose-Response Curve will be generated for mean time to nodal and visceral progressions at different dose level
Dose response relationship within setting of re-irradiation (infield progressions) | From date of start of treatment of disease progression, assessed upto 3 years
  Radiation Dose-Response Curve will be generated for mean time to infield progression at different dose level
Moderate to severe adverse events within the (induced) oligo-metastatic and oligo-recurrent setting ( including toxicity with targeted agents like bevacuzimab and pembrolizumab) | From date of start of treatment of recurrence to end of study, assessed upto 3 years after initiation of the study
  Number or percent of participants with treatment-related moderate to severe adverse events as assessed by CTCAE v4.0 (If available)
Report on various risk groups within oligo-metastatic and oligo-recurrent setting | From date of recurrence to end of study, assessed upto 3 years after initiation of the study
  Clinical, pathological, and treatment-related factors of patients recorded during the sudy will be used to develop multivariable risk models to identify risk factors and define various risk groups within oligo-metastatic and oligo-recurrent setting
Nomogram which correlates risk groups with expected outcomes within the (induced) oligo-metastatic and oligo-recurrent setting | From date of recurrence to end of study, assessed upto 3 years after initiation of the study
  Nomogram will be developed which could estimate the probability of a expected outcomes (overall survival, infield progression free survival, overall progression free survival) based on the risk group the patient belongs to within oligo-metastatic and oligo-recurrent setting.
Tissue based biomarkers | From date of start of recurrence to end of study, assessed upto 3 years after initiation of the study
  Sponsor Institute will facilitate storage of biopsy tissue of patients within oligo-metastatic and oligo-recurrent setting included in this study. In future, these tissue samples will be used for translational reseach in this field.

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Chopra, MD, DNB, Principal Investigator — Tata Memorial Centre; Remi A Nout, MD, Phd, Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: Undecided